CLINICAL TRIAL: NCT04753788
Title: Clinical Evaluation of a Loop-mediated Isothermal Amplification Test for Treponema Pallidum Pertenue: A Diagnostic Tool to Support Yaws Eradication
Brief Title: Evaluation of a LAMP Assay for T. Pallidum. Pertenue
Acronym: LAMP4YAWS
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Pasteur Institute abidjan (Unknown); Centre Pasteur du Cameroun (Other); Noguchi Memorial Institute for Medical Research (Other); University of Freiburg (Other); MAST Group - Germany (Unknown); Friedrich-Loeffler-Institut (Unknown); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Other Study IDs: LSHTM-21633
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Yaws
MeSH Terms: conditions — Yaws

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Yaws Cases: Individuals with a lesion clinically suspected to be yaws and with evidence of positive treponemal and non-treponemal serology as assessed by point of care lateral flow tests (DPP Syphilis Screen and Confirm, Chembio)
  Interventions: Diagnostic Test: PCR; Diagnostic Test: LAMP

INTERVENTIONS:
Diagnostic Test: PCR — qPCR for T.pallidum
Diagnostic Test: LAMP — LAMP assay for T.pallidum

SUMMARY:
This is a diagnostic evaluation comparing the performance of real-time PCR performed at a national reference laboratory and a LAMP assay performed at a regional hospital for the diagnosis of yaws

ELIGIBILITY:
Inclusion Criteria:

* Lesion consistent with yaws
* Positive treponemal and non-treponemal antibodies assessed by the DPP Syphilis Screen and Confirm RDT

Exclusion Criteria:

* Unable to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with clinically suspected yaws lesions in Ghana, Cote d'Ivoire and Cameroon will be screened using the DPP Syphilis Screen and Confirm RDT. If positive samples will be taken for PCR and LAMP testing.
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Centre Pasteur, Yaoundé, Cameroon
- Institut Pasteur, Abidjan, Côte d’Ivoire
- Noguchi Memorial Institute of Medical Research, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Handley BL, Gonzalez-Beiras C, Tchatchouang S, Basing LA, Hugues KA, Bakheit M, Becherer L, Ries C, Njih Tabah E, Crucitti T, Borst N, Luert S, Frischmann S, Haerpfer T, Landmann E, Amanor I, Sylla A, Kouame-Sina MS, Ndzomo-Ngono JP, Tano A, Arhinful D, Awondo P, Ngazoa Kakou S, Eyangoh S, Addo KK, Harding-Esch EM, Knauf S, Mitja O, Marks M. LAMP4yaws: Treponema pallidum, Haemophilus ducreyi loop mediated isothermal amplification - protocol for a cross-sectional, observational, diagnostic accuracy study. BMJ Open. 2022 Mar 29;12(3):e058605. doi: 10.1136/bmjopen-2021-058605. PMID 35351731

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suspected Yaws Cases
Started | 563
Completed | 525 (7 individuals without an RNAseP result and 31 missing either LAMP or qPCR)
Not Completed | 38

BASELINE CHARACTERISTICS:
Arm/Group | Suspected Yaws Cases
Number analyzed (Participants) | 525
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 525
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 376
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 525
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Cameroon | 20
  Côte D'Ivoire | 93
  Ghana | 408
  Congo | 4

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of LAMP vs qpCR
Description: A case of Yaws Positive for T.pallidum DNA by PCR that is also positive by LAMP
Time Frame: 15 Months
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- Serologically Confirmed Yaws: Positive serological test for yaws
Arm/Group | Serologically Confirmed Yaws
Number analyzed (Participants) | 525
Percent | 63.2 [60.6 to 70.9]

2. Primary Outcome: Specificity of LAMP for Yaws
Description: Sample negative by qPCR for T.pallidum that is also negative by LAMP
Time Frame: 15 Months
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Serologically Confirmed Yaws
Number analyzed (Participants) | 525
Percent | 67.1 [61.6 to 72.8]

ADVERSE EVENTS:
Time Frame: This is a diagnostic accuracy study without collection of data on AE/SAEs
Description: This is a diagnostic accuracy study without collection of data on AE/SAEs
Arm/Group | Suspected Yaws Cases
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04753788/Prot_SAP_000.pdf